CLINICAL TRIAL: NCT00860288
Title: Efficacy and Long-Term Safety of Vildagliptin as Add-on Therapy to Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237B2224
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Vildagliptin Dose 1 (Experimental)
  Interventions: Drug: Vildagliptin; Drug: Metformin
- Vildagliptin Dose 2 (Experimental)
  Interventions: Drug: Vildagliptin; Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Metformin; Drug: Placebo
- Sitagliptin (Active Comparator)
  Interventions: Drug: Metformin; Drug: Sitagliptin

INTERVENTIONS:
Drug: Vildagliptin
  Arms: Vildagliptin Dose 1; Vildagliptin Dose 2
Drug: Metformin
Drug: Placebo
  Arms: Placebo
Drug: Sitagliptin
  Arms: Sitagliptin

SUMMARY:
This is a 2-3 period parallel group study with an adaptive element in Type 2 diabetes patients receiving vildagliptin as add-on therapy to metformin

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-78 years old inclusive at Visit 1
* T2DM patients treated with metformin for at least 3 months and a stable dose of at least 1500 mg daily for a minimum of 4 weeks prior to Visit 1
* Patient agreement to maintain same dose of metformin throughout study
* HbA1c of ≥ 7.0 and ≤ 9.5 % at Visit 1
* Body Mass Index (BMI) in the range of 22-45 kg/m2 at visit 1

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* FPG ≥ 270 mg/dL ( ≥ 15.0 mmol/L)

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1988 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of vildagliptin as add-on therapy to metformin in patients with T2DM by assessing changes in HbA1c with vildagliptin added to metformin to that of placebo added to metformin after 24 weeks of treatment | 24 weeks

SECONDARY OUTCOMES:
To evaluate the efficacy of vildagliptin as add-on therapy to metformin in patients with T2DM by assessing changes in HbA1c with vildagliptin added to metformin to that of sitagliptin added to metformin after 24 weeks of treatment. | 24 weeks
To evaluate the efficacy of vildagliptin as add-on therapy to metformin in patients with T2DM by assessing changes in fasting plasma glucose with vildagliptin added to metformin to that of placebo added to metformin after 24 weeks of treatment. | 24 weeks
To evaluate the efficacy of vildagliptin as add-on therapy to metformin in patients with T2DM by assessing changes in fasting plasma glucose with vildagliptin added to metformin to that of sitagliptin added to metformin. | 24 weeks
To evaluate the safety and tolerability of vildagliptin compared to placebo and sitagliptin over 24 weeks of treatment as add-on therapy to metformin in patients with T2DM. | 24 weeks
To evaluate the long-term safety and tolerability of vildagliptin compared to sitagliptin over the entire study duration as add-on therapy to metformin in patients with T2DM. | 76 weeks
To evaluate the body weight change from baseline with vildagliptin compared to placebo and sitagliptin after 24 weeks of treatment as add-on therapy to metformin in patients with T2DM. | 24 weeks
To evaluate the long-term efficacy of vildagliptin compared to sitagliptin over the entire study duration as add-on therapy to metformin in patients with T2DM. | 76 weeks

CONTACTS AND LOCATIONS:
Locations (185):
- Argentina (6):
  - Instituto de Investigaciones Biomedicas, Buenos Aires, Santa Fe Province
  - Grupo Colaborative Rosario, Rosario, Santa Fe Province
  - Grupo Medico Alem, Buenos Aires
  - DIM Clinical Privada, Buenos Aires
  - Clinica Medica Sin Internacion, Buenos Aires
  - Fundación de Estudios Farmacológicos y de Medicamentos, Buenos Aires
- Austria (5):
  - Universitaetsklinik Graz medizinische Universitaetsklinik;, Graz
  - LKH Salzburg Landesklinik fuer Innere Medizin I, Salzburg
  - Millergasse 7, Vienna
  - Hanusch Krankenhaus 1. Med. Abteilung und Nephrodepartment, Vienna
  - Kindlergasse 4, Wiener Neustadt
- Belgium (6):
  - Private Practice Diabetology (Dr. Coucke), Sint-Gillis-Waas, Sint-Niklaasstraat 117
  - Private Practice Cardiology (Dr. Hollanders), De Pinte
  - Private Practice (Vernijns), Genk
  - Private Practice (Dr. De Meulemeester), Gozée
  - Huisartsenpraktijk Hygeia, Hasselt
  - Private Practice (Dr. Jaak Mortelmans), Oostham
- Finland (8):
  - Lihavuustutkimusyksikkö, Helsinki
  - Mehiläinen Töölö Diabetesklinikka, Helsinki
  - Terveystalo Kuopio, Kuopio
  - Mehiläinen Lahti, Lahti
  - ODL Terveys Oy, Tutkimusyksikkö,, Oulu
  - Mehiläinen Riihimäki, Riihimäki
  - Terveystalo Tampereen työterveys Kalmar, Tampere
  - Myyrmäen terveysasema, Vantaa
- Germany (51):
  - Internistische Gemeinschaftspraxis Nagel, Dietlein & Hunstiger, Augsburg
  - Praxis Dr. Med. Kurt Rack, Augsburg
  - Gemeinschaftspraxis S. Maxeiner/Dr. Behr/S. Rupprecht, Bad Kreuznach
  - Klinische Forschung Berlin-Buch, Berlin
  - Praxis Dr. Med. Ulrike Venschott-Jordan, Berlin
  - Praxis Dr. Med. Monika Kiper, Berlin
  - Praxis Dr. Med. Christina Bondke, Berlin
  - Bibertal Klinik, Bibertal
  - Praxis Dr. Med. Claudia Ulbrich, Cologne
  - Gemeinschaftspraxis Dr. med. Ali Boustani, Diez
  - Facharzt fuer Allgemeinmedizin, Dorsten
  - Praxis Dr. Med. Anwar Ansari, Einbeck
  - Hausaerzte am Stern Dr. Med. Blume / Dr. Med. Garanin, Essen
  - Praxis Dr. Med. Roland Kutzke, Essen
  - Praxis Dr. Med. Thorsten Rau, Essen
  - Praxis Dr. Med. Joerg Luedemann / Facharzt fuer Innere Medizin - Diabetologie, Falkensee
  - Praxis Dr. Med. Daniela Freise, Frankfurt
  - Dial.-Med. Kerstin Steinbach, Freital
  - Gemeinschaftspraxis, Fulda
  - Praxis Dr. Med. Wolfgang Krause, Grimma
  - Krankenhaus Hagenow, Innere Medizin, Hagenow
  - MVZ-medicum Hamburg, Hamburg
  - Diabetes-Zentrum Wandsbek, Hamburg
  - Gemeinschaftspraxis Dr. Grüneberg, Dr.Mehring, Bitterer-Tölle, Herne
  - Praxis Dr. Med. Helmut Anderten, Hildesheim
  - Praxis Dr. Med. Juergen Landschulze, Kahla
  - Praxis Dr. Med. Julia Chevts, Karlsruhe
  - Praxis Dr. Med. Hans-Helmut Seibert, Kassel
  - Dres. Klein/Minnich, Künzing
  - Praxis Dr. Med. Birgit Hoene, Leipzig
  - Pro Scientia med, Lübeck
  - Diabetes Schwerpunktpraxis, Meissen
  - Praxis Dres. Prohaska / Lindner, Mühldorf
  - Praxis Dr. Med. Claus-Michael Grimm, München
  - Praxis Dr. Fischer & Dr. Keuthage, Münster
  - Gemeinschaftspraxis Dr. Uwe Böckmann/Dr. med. Maren Molkewehrum, Neumünster
  - Praxis Dr. Med. Joachim Etter, Oberhausen
  - IkFE Studiencenter Potsdam GMBH i.G., Potsdam
  - Diabetes Center Quakenbrueck, Quakenbrück
  - Praxis Dr. Altwicker, Dr. Kanis, Reinfeld
  - Praxis Dr. Med. Ulrich Aigner, Rothenburg
  - Praxis Dr. Med. Sabine Sedl, Schönberg
  - Dres. Hiltensperger & Schaal, Schrobenhausen
  - Praxis Hans-Joachim Herrmann/Dr. med. B. Bauer, Schwabenheim
  - Praxis Dr. Med. Ottmar Herfert, Stuttgart
  - Praxis Dr. Med. Doru Popa, Veitsbronn
  - Gemeinschaftspraxis Gerhard Steinmaier und Dr. Med. Werner Bauer, Viernheim
  - Gemeinschaftspraxis Sauter, Wangen
  - Praxis Dr. Med. Rudolf Matthias Remppis, Weißenhorn
  - Praxis Dr. Med. Peter Genthner, Welzheim
  - Gemeinschaftspraxis Dr. med. Reinhold Schneider und Christine Schneider, Wetzlar
- Greece (3):
  - Laiko General Hospital,, Athens
  - Lamia General Hospital, Larissa
  - Papageorgiou General Hospital, Thessaloniki
- Guatemala (5):
  - Clínica y Hospital Colón del Paciente Diabético, Guatemala City
  - Endonutri S.A, Guatemala City
  - Clinica Dr. Erick Turcios, Guatemala City
  - Endonutri S. A., Guatemala City
  - Clinica Dr. Sergio Bran, Guatemala City
- Hungary (9):
  - Szent Margit Hospita, Budapest
  - Károlyi Sándor Hospital, Budapest
  - Szent Imre Hospital, Budapest
  - Konszenzusplusz Kft., Csongrád
  - Petz Aladar Hospital, Győr
  - Jósa Andras Hospital, Nyíregyháza
  - Szte-Áok I, Szeged
  - Balassa Janos Hospital, Szekszárd
  - Zala Megyei Hospital, Zalaegerszeg
- India (9):
  - Manipal Hospital,, Bangalore, Karantaka
  - Health and Research Centre, Trivandrum, Kerala
  - Diabetes Thyroid Hormone Research Institute Pvt Ltd., Indore, Madhya Pradesh
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - M. V. Hosp for Diabetes P. Ltd. 4,, Chennai
  - Medicity Hospital, Hyderabaad
  - Nizam's institute of medical sciences,, Hyderabaad
  - S. R. Kalla Memorial gastro and general hosp,, Jaipur
  - Christian Medical College,, Vellore
- Israel (2):
  - Maccabi Healthcare Services, Rishon LeZiyyon
  - Ziv Medical Center, Safed
- Italy (20):
  - U.O.C. di Diabetologia e Malattie Metaboliche, Arenzano
  - U.S.C. di Endocrinologia (Ingresso 13 - piano 2) Dip. di Medicina, Bergamo
  - U.O.C. Diabetologia Endocrinologia Dip. Medico, Campobasso
  - U.O. Medicina Generale, Casorate Primo
  - I Divisione Medicina, Catania
  - U.O. Malattie Metaboliche e Diabetologia, Chieri
  - U.O.C. di Medicina d'Urgenza e Pronto Soccorso, Cosenza
  - Servizio Diabetologia, SOD Cardiologia Geriatrica - D.A.I. del Cuore e dei Vasi, Florence
  - Centro Diabetologico Malattie Metaboliche, Mercato San Severino
  - Divisione Malattie Metaboliche e Diabetologia, Milan
  - S. Semplice Dip. di Endocrinologia e Diabetologia Dip. di Medicina Interna, Milan
  - U.O. Medicina II - Dip. Medicina Interna, Milan
  - Unità Cardio-Metabolica e Trials Clinici Dipartimento di Medicina Interna, Milan
  - U.O. Diabetologia, Olbia
  - Centro per l'Aterosclerosi Dip. di Medicina Interna, Roma
  - U.O. Endocrinologia e Diabetologia, Roma
  - U.O.C. di Diabetologia c/o AUSL ROMA B - Sede Territoriale, Roma
  - U.O.C. di Medicina Interna B - BMI02 Dip. Scienze Cliniche - II Clinica Medica, Roma
  - S. S. di Diabetologia Dip. Med. Interna e Malattie Metaboliche, Siena
  - S.C. Prevenzione-Riabilitazione Cardiologica presso ex-Dispensario, Vibo Valentia
- Latvia (7):
  - Daugavpils Regional Hospital, Daugavpils
  - Primary Health Centre of Jaunliepaja, Liepāja
  - Private practice of endocrinology, Ogre
  - Center of Endocrinology, Riga
  - Riga Outpatient Clinic "Dziednieciba", Riga
  - Talsi Clinical Hospital, Talsi
  - Endocrinology Department of Vidzemes Hospital, Valmiera
- Lithuania (7):
  - JSC "Klinikiniai sprendimai", Alytus
  - Kaunas District Hospital, Kaunas
  - Kaunas Silainiai Outpatient Clinic, Kaunas
  - Kaunas Medical University Hospital, Kaunas
  - Kaunas Dainavos Outpatient Clinic, Kaunas
  - Vilnius University Hospital Santariskiu Clinics, Vilnius
  - Private Endocrinology Clinic, Vilnius
- Mexico (5):
  - Comité Bioetico para la Investigación Clínica S.C., Mexico City, Durango
  - Unidad Metabolica y Cardiovascular S.C., Cuernavaca, Morelos
  - Clínica Eugenio Sue, Mexico City, Polanco Chapultepec
  - Clínica de Diabetes de la Secretaria de Salud de Durango, Durango
  - Arke Estudios Clinicos S.A. de C.V., Mexico City
- Norway (6):
  - Flattum legesenter, Hønefoss
  - Randesund Helsesenter, Kristiansand
  - Sinsenklinikken, Oslo
  - Oslo Universitetssykehus, Oslo
  - Hinnastrekanten legekontor, Stavanger
  - Vennesla legesenter, Vennesla
- Peru (6):
  - Clinica San Miguel, Arequipa
  - Clinica Geriatrica Militar, Lima
  - Clinica San Borja, Lima
  - Clinica Senor de los Milagros, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
- Poland (5):
  - Bydgoskie Centrum Diabetologii i Endokrynologii, Bydgoszcz
  - NZOZ "Specjalista" Sp z o. o., Kutno
  - Oddzial Chorob Wewnetrznych, Mielec
  - Poradnia Lekarza Rodzinnego, Poznan
  - Poznański Ośrodek Medyczny "NOVAMED", Poznan
- Romania (7):
  - CMI Cardiologie "Dr. Pop Calin Florin", Baia Mare
  - "C. I. Parhon" Endocrinology Institute, Bucharest
  - Medical Centre "Sanatatea Ta" SRL, Bucharest
  - Medical Practice SRL, Oradea
  - Anamed SRL, Oradea
  - Emergency County Hospital Ploiesti, Ploieşti
  - Policlinica "Dr. Citu", Timișoara
- Slovakia (10):
  - MEDISPEKTRUM s.r.o,, Bratislava, Slovak Republic
  - .Interna klinika, FN J.A. Reimana, Prešov, Slovak Republic
  - Diabetologicka ambulancia,, Bratislava, Slovakia Republic
  - Diabetologicka ambulancia, Košice, Slovakia Republic
  - Diabetologicka ambulancia,, Lučenec, Slovakia Republic
  - NZZ Diabetologicka ambulancia, Nové Zámky, Slovakia Republic
  - Diabetes centrum s.r.o, Trenčín, Slovakia Republic
  - Diabetologicka ambulancia,, Žilina, Slovakia Republic
  - Diametabol.s.r.o.,, Bratislava
  - MUDr. Margita Kiripolska s.r.o, Považská Bystrica
- South Korea (5):
  - Eulji General Hospital, Seoul
  - Kangbuk Samsung Medical center, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea Holy Family Hospital, Seoul
  - Ajou university hospital, Suwon
- Venezuela (3):
  - Ambulatorio Militar Tipo III Paramacay. Avenida Universidad. Sector Santa Ana. Naguanagua., Valencia, Carabobo
  - Hospital Militar Dr Carlos Arvelo. Final Av. José Angel Lamas. Servicio de Endocrinología., Caracas
  - Hospital Dr Miguel Perez Carreño. Servicio de Endocrinología. Sotano., Caracas

REFERENCES:
- See also: Results for CLAF237B2224 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5663